CLINICAL TRIAL: NCT05374291
Title: A Randomized Controlled Clinical Trial to Assess the Effect of Dapagliflozin on Renal and Cardiovascular Outcomes in Patients With Severe Chronic Kidney Disease
Brief Title: The RENAL LIFECYCLE Trial: A RCT to Assess the Effect of Dapagliflozin on Renal and Cardiovascular Outcomes in Patients With Severe CKD
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: AstraZeneca (Industry); Dutch Kidney Foundation (Other)
Responsible Party: Principal Investigator, Ron Gansevoort, prof. dr. R.T. Gansevoort, MD PhD, FERA, FASN, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202100617; 2021-005446-15 (EudraCT Number); 2023-508389-13-00 (EU CTIS Number)
Record Dates: First submitted 2022-04-22; First posted 2022-05-16 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Kidney Disease, Chronic; Renal Transplant Failure; Heart Failure; Kidney Failure; Death
Keywords: advanced CKD; dialysis; kidney transplant; all-cause mortality; kidney failure; hospitalization for heart failure; Dapagliflozin
MeSH Terms: conditions — Renal Insufficiency, Chronic; Heart Failure; Renal Insufficiency; Death | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: The RENAL LIFECYCLE trial consists of a screening period and a double blind treatment period with two arms. Participants will be randomly assigned in a 1:1 ratio to double blind treatment with dapagliflozin 10 mg/d or matching placebo. Randomization will be stratified by enrolment stratum (pre-dialysis, dialysis, kidney transplantation), centre and type 2 diabetes mellitus status yes/no) to ensure balanced distribution across the two treatment arms.
Who Masked: Participant, Investigator
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin 10 mg/day (oral)
  Interventions: Drug: Dapagliflozin 10 mg/day (oral)
- Placebo (Placebo Comparator): Placebo 10 mg/day (oral)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10 mg/day (oral) — Patients take 10 mg dapagliflozin or matching placebo once daily in the morning
  Other Names: Forxiga
  Arms: Dapagliflozin
Drug: Placebo — Patients take 10 mg dapagliflozin or matching placebo once daily in the morning
  Arms: Placebo

SUMMARY:
Rationale:

Sodium glucose co transporter 2 (SGLT2) inhibitors are a relatively new class of agents, originally developed as oral antihyperglycemic drugs. SGLT2 inhibitors are clinically available since 2012 for the treatment of patients with diabetes mellitus type 2. Later, SGLT2 inhibitors appeared to have also specific reno- and cardioprotective effects. Remarkably, the trials that have been performed thus far excluded patients with an eGFR below 25 mL/min/1.73m2 at inclusion, prevalent dialysis patients, and kidney transplant recipients. This is unfortunate, because especially these patients are at high risk of reaching kidney failure requiring dialysis, cardiovascular complications and mortality, whereas there are only few proven effective therapies. There is emerging evidence from experimental studies and post hoc-analyses of randomized clinical trials that SGLT2 inhibitors may also be effective in preventing cardiovascular and mortality outcomes in these patients with severe CKD, including patients receiving dialysis or living with a kidney transplant. For instance, subgroup analysis of the DAPA-CKD trial comparing 624 patients with an eGFR<30 to the remainder of the trial population with better kidney function, demonstrated that the efficacy of the SGLT2 inhibitor dapagliflozin in reducing cardiovascular, heart failure and renal outcomes persisted in the population with impaired kidney function. Furthermore, in the DAPA-CKD trial patients continued to use dapagliflozin or placebo when dialysis was initiated. In the subgroup of patients who initiated dialysis, dapagliflozin was associated with a relative risk reduction for mortality of 21%. Finally, in kidney transplant recipients, SGLT2 inhibitors have been shown to be effective in lowering HbA1c, body weight, blood pressure and stabilize kidney function, and these agents were well tolerated and safe. Taken these findings together there is a sound rationale to study the long-term reno- and cardioprotective efficacy and safety of SGLT2 inhibitors in patients with severe CKD.

There are two cardiac sub-studies: the cardiac magnetic resonance imaging (MRI) sub-study and the echocardiography sub-study. The echocardiography sub-study is referred to as the "SGLT-2-inhibitors to Target Heart Failure in Peritoneal Dialysis" (STOP-HF-in-PD) study.

DETAILED DESCRIPTION:
Objective:

To establish the reno- and cardioprotective efficacy and safety of dapagliflozin in patients with severe CKD

Study design:

Multicenter, randomized, controlled, double blinded, pragmatic, interventional trial

Study population:

* Patients with advanced CKD, i.e. an eGFR ≤25 mL/min*1.73m2
* Patients on dialysis (at least 3 months after start of dialysis)
* Patients with a kidney transplant and an eGFR ≤45 mL/min/1.73m2 (at least 6 months after transplantation)

Intervention:

Dapagliflozin 10 mg/day or matching placebo

Primary outcome measure:

Combined endpoint of all-cause mortality, kidney failure, and hospitalization for heart failure in the overall study population

Study duration:

18 month recruitment phase, 30 month follow-up after enrollment of the last patient: Total study duration intended to last 48 months. It should be noted that the trial is event driven and will be terminated when 468 primary composite outcomes have occurred. The exact trial duration may therefore be shorter or longer than the intended 48 months.

Study visits:

Screening, baseline, week 2, month 3, month 6 and every 6 months thereafter. Information needed for the trial will be obtained as much as possible from visits taking place as part of routine clinical care.

Sample size:

Renal Lifecycle is designed as an endpoint driven trial and will finish when 468 primary study outcomes have occurred. The investigators have estimated a sample size of 1750-2000 patients.

Novel aspects:

A unique patient population with severe chronic kidney disease at very high risk of adverse outcomes for whom very few proven effective therapies exist. The initiation and efficacy of SGLT2 inhibitors, including dapagliflozin, has not been studied before in this population. However, SGLT2 inhibitors have the potential to be very effective and well tolerated which would imply a major advance in the pharmacotherapy of these patients.

When patients reach a renal endpoint, e.g. start or chronic dialysis or receiving a kidney transplantation, study medication will not be stopped as customary in many other trials in nephrology, but continued in the new phase of their "renal lifecycle", hence the name of the trial.

Sub studies:

Cardiac MRI sub-study The cardiac MRI sub-study will evaluate the effect of dapagliflozin on cardiac remodelling, as compared to placebo, measured with indexed left ventricular mass (LVMi), an intermediate cardiovascular outcome, in 250 participants across all three groups of the Renal Lifecycle Trial (i.e. advanced CKD, dialysis, kidney transplant recipients). This will provide robust evidence on the mechanisms under-pinning the cardioprotective effects of SGLT2 inhibitors in this high-risk patient population.

Primary outcome: Difference in LVMi after 12 months dapagliflozin compared to placebo.

Secondary outcomes: Differences between intervention groups in the following parameters at 12 months post-randomization: non-indexed LVM; indexed left atrial volume; non-indexed left atrial volume; indexed left and right ventricular end diastolic volume; indexed left and right ventricular end systolic volume; left and right ejection fraction.

Echocardiography sub-study (STOP-HF-in-PD) The echocardiography sub-study (STOP-HF-in-PD) will evaluate the effect of dapagliflozin on cardiac function, as compared to placebo, measured by left ventricular global longitudinal strain (LV-GLS), in 100 participants with kidney failure treated with peritoneal dialysis (PD). This will provide additional evidence on the mechanisms underlying the cardiac effects of SGLT2i in patients with kidney failure. Furthermore, the LV-GLS-data will be related to measured CKD- and PD-associated mediators of heart failure (measured in serum, urine and peritoneal effluent). This will aid to determine their relevance in patients with kidney failure, as well as to define if and to what extent SGLT2i affect these mediators in patients with kidney failure.

Primary outcome: Difference in LV-GLS after 6 months dapagliflozin compared to placebo.

Secondary and exploratory objectives: Differences between dapagliflozin compared to placebo after 6 and 12 months post-randomization for: LV-GLS; E/e'-ratio; left atrial volume index; left atrial strain; tricuspid velocity; left ventricular ejection fraction; LVMi; Physical functioning (6 minute walking test and KCCQ-12); 24h urine volume; residual kidney function; average daily ultrafiltration volume; peritoneal glucose exposure; peritoneal membrane characteristics.

Combined Cardiac Imaging Sub-studies A subset of participants enrolled in the echocardiography sub-study will also participate in the cardiac MRI sub-study, allowing for a combined evaluation of both imaging modalities. The aim is to evaluate the use of echocardiography and cardiac MRI as a tool to identify patients at highest risk for heart failure and those who may benefit from SGLT2i-induced cardio-protection.

Secondary outcomes: Association between change in LV-GLS and change in LVMi from baseline to 12-months across intervention groups; association between change in LV-GLS at 6 months and change in LVMi at 12 months across intervention groups.

Cognitive sub-study Patients with chronic kidney disease (CKD) are at a much higher risk for developing cognitive impairment compared with the general population and both lower glomerular filtration rate and the presence of albuminuria are associated with its development. SGLT-2 inhibitor use is associated with better preservation of cognitive function in patients with CKD including those on hemodialysis and after kidney transplantation compared to placebo.Patients will be requested to perform the symbol digit modalities test at the same time as the questionnaires, i.e. at baseline (visit 2), visit 5 and visit 6, once every year after visit 6 and at EoT/EET.The primary outcome of the cognition sub study is the change over time in the number of correct answers in the symbol digit modalities test within 90 seconds.

Kidney metabolism substudy The primary aim of this substudy is to evaluate the effect of dapagliflozin 10 mg compared to a placebo on energy metabolism assessed by changes in the renal mitochondrial oxidative phosphorylation capacity in kidney transplant recipients participating in the RENAL LIFECYCLE Trial at the 3-month Follow-up Visit. Further aims of this substudy are to evaluate the differences in metabolic substrate preferences by measuring ketone body or acylcarnitine substrate-driven mitochondrial respiration following the randomization to dapagliflozin or placebo.

Differences in mitochondrial architecture including mitochondrial quantity and morphology will be assessed using electron microscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced CKD i.e. an eGFR ≤25 mL/min/1.73m2
* Dialysis patients (at least 3 months after start of dialysis)
* Transplant patients with an eGFR ≤45 mL/min/1.73m2 (at least 6 months after transplantation)

In addition, to be eligible all subjects must meet all criteria below

* Age >18 years
* Willing to sign informed consent
* Pre-dialysis patients with eGFR ≤25 mL/min/1.73m2 have to be on a stable dose (no changes in dose or type of drug) of ACEis or ARBs for at least 4 weeks prior to the screening visit to be eligible to proceed to the randomization visit unless there is documented evidence that the patient does not tolerate an ACEi or ARB. These subjects will maintain their stable doses of ACEis or ARBs throughout the trial (when possible and tolerated by the patient). ACEi or ARBs are not required for patients on maintenance dialysis or kidney transplant recipients.

Exclusion Criteria:

* Mentally incapacitated subjects (i.e. not able to sign informed consent)
* Diagnosis of type 1 diabetes mellitus
* Concurrent treatment with SGLT2 inhibitor
* History of ≥2 urinary tract / genital infections during the last six months
* Life expectancy <6 months in the opinion of the treating physician.
* Scheduled start of dialysis within 3 months or kidney transplantation within 6 months
* patients treated for a renal indication during the last 6 months with a course of systemic immunosuppressive agents or intensification of treatment with systemic immunosuppressive agents, such as patients with a kidney transplant and acute rejection or patients with GPA (Morbus Wegener) and a recent flare.
* Active malignancy aside from treated squamous cell or basal cell carcinoma of the skin.
* History of severe hypersensitivity or known severe hepatic impairment (Child-Pugh class C)
* History of severe noncompliance to medical regimens or unwillingness to comply with the study protocol.
* Pregnancy or breastfeeding
* Presence of other transplanted organ besides a kidney transplant
* Severe lactose intolerance
* Autosomal Dominant Polycystic Kidney Disease (ADPKD) treated with tolvaptan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1750 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of partipants with all-cause mortality, kidney failure, and hospitalization for heart failure | Total study duration intended to last 48 months
  To determine whether dapagliflozin is superior to placebo in reducing the incidence of the primary composite endpoint
  Combined endpoint of all-cause mortality, kidney failure, and hospitalization for heart failure in the overall study population

SECONDARY OUTCOMES:
Number of participants to reach all-cause mortality | Total study duration intended to last 48 months
  To determine if dapagliflozin is superior to placebo in reducing the incidence of all-cause mortality
Incidence of hospitalization for heart failure | Total study duration intended to last 48 months
  Incidence of hospitalization for heart failureTo determine if dapagliflozin is superior to placebo in reducing the incidence of heart failure
Incidence of kidney failure (chronic dialysis, kidney transplantation or mortality due to kidney failure) | Total study duration intended to last 48 months
  To determine if dapagliflozin is superior to placebo in reducing the incidence of kidney failure
incidence of the composite outcome (kidney failure, hospitalization for heart failure, and all-cause mortality) in subgroups | Total study duration intended to last 48 months
  To determine whether dapagliflozin is superior to placebo in reducing the incidence of the composite outcome in subgroups
  subgroups: advanced CKD i.e. an eGFR ≤30 mL/min/1.73m2, dialysis patients and transplant patients

OTHER OUTCOMES:
measuring Quality of life with the EQ-5D questionnaire | Total study duration intended to last 48 months
  To determine whether dapagliflozin is superior to placebo in comparing the Quality of Life for all subgroups based on the EQ-5D questionnaire
measuring Quality of life with the SF12 questionnaire | Total study duration intended to last 48 months
  To determine whether dapagliflozin is superior to placebo in comparing the Quality of Life for all subgroups based onthe SF12 questionnaire
Cost-effectiveness of SGLT2-inhibition using the Quality of Life-data derived from the EQ-5D and SF-12 questionnaires | Total study duration intended to last 48 months
  cost-effectiveness of SGLT2-inhibition in the overall study population as well as in the three subpopulations
incidence of de-novo type 2 diabetes in patients without diabetes | Total study duration intended to last 48 months
  To determine whether dapagliflozin is superior to placebo in reducing the incidence of de-novo type 2 diabetes
Change in the eGFR slope | Total study duration intended to last 48 months
  To determine whether dapagliflozin is superior to placebo in reducing the eGFR slope
  eGFR slope; for the dialysis subgroup slope residual kidney function will be calculated using the average of 24hr urinary creatinine and urea clearance values over time
incidence of diuresis <200 ml/24hr in the dialysis subgroup | Total study duration intended to last 48 months
  To determine whether dapagliflozin is superior to placebo in the incidence of diuresis <200 ml/24hr in the dialysis subgroup
  for this purpose 24hr urine samples will be collected ≥2 times per year
incidence of the composite outcome (kidney failure, hospitalization for heart failure, and all-cause mortality) in subgroups with and without type 2 diabetes separately | Total study duration intended to last 48 months
  To determine if dapagliflozin is superior to placebo in reducing the incidence of kidney failure with and without type 2 diabetes separately

CONTACTS AND LOCATIONS:
Overall Officials: Ron Gansevoort, Principal Investigator — University Medical Center Groningen
Locations (90):
- Australia (18):
  - Canberra Health Services, Canberra, Australian Capital Teritory
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Concord Repatriation General Hospital, Sydney, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - St George Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Sunshine Coast Hospital and Health Services, Birtinya, Queensland
  - Royal Brisbane and Womens Hospital, Brisbane, Queensland
  - Townsville University hospital, Douglas, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Western Health, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - East Metro Health Services (Royal Perth Hospital and Armadale Health Services), Perth, Western Australia
  - Box Hill Hospital (Eastern Health), Melbourne
- Belgium (4):
  - UZ Brussel, Brussels
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - AZ Glorieux, Ronse
- Germany (17):
  - Charité, Berlin
  - Praxis für Dialyse und Nierenkrankheiten, Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Halle (Saale) Innere Medizin 2, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Zentrum fuer Nieren-, Hochdruck- und Stoffwechselerkrankungen Hannover, Hanover
  - Nierenzentrum Heidelberg, Heidelberg
  - Dialysezentrum Heilbronn - Überörtliche Berufsausübungsgemeinschaft für Nephro und Dialyse (ÜBAG), Heilbronn
  - Universitätsklinikum JenaKlinik für Innere Medizin III, Jena
  - Universitätsmedizin Mainz, Mainz
  - Universitätsklinikum RegensburgAbteilung für Nephrologie, Regensburg
  - Universitätsklinikum Tübingen Medizinische Klinik IV, Tübingen
  - Universitätsklinikum Ulm, Klinik für Innere Medizin I, Nephrologie, Ulm
  - Nephrologisches Zentrum Villingen/Schwenningen, Villingen-Schwenningen
  - Nierenzentrum Wiesbaden, Wiesbaden
  - Medizinische Klinik und Poliklinik I der Universitätsklinik WürzburgSchwerpunkt Nephrologie, Würzburg
- Netherlands (45):
  - Wilhelmina Ziekenhuis Assen, Assen, Drenthe
  - Flevoziekenhuis, Almere Stad, Flevoland
  - Gelre Ziekenhuizen, Apeldoorn, Gelderland
  - Laurentius Ziekenhuis, Roermond, Limburg
  - Zuyderland Medisch Centrum, Sittard, Limburg
  - Amphia Ziekenhuis, Breda, North Brabant
  - Amsterdam UMC, Amsterdam, North Holland
  - OLVG, Amsterdam, North Holland
  - Ziekenhuisgroep Twente, Almelo, Overijssel
  - Saxenburgh Medisch Centrum, Hardenberg, Overijssel
  - Dialyse Centrum Groningen, Groningen, Provincie Groningen
  - UMCG, Groningen, Provincie Groningen
  - Albert Schweitzer ziekenhuis, Dordrecht, South Holland
  - Alrijne, Leiderdorp, South Holland
  - Erasmus Medisch Centrum, Rotterdam, South Holland
  - Maasstad Ziekenhuis, Rotterdam, South Holland
  - Haaglanden Medisch Centrum, The Hague, South Holland
  - HagaZiekenhuis, The Hague, South Holland
  - Admiraal de Ruyter Ziekenhuis, Goes, Zeeland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Noordwest Ziekenhuisgroep Alkmaar, Alkmaar
  - Meander Medisch Centrum, Amersfoort
  - Niercentrum aan de Amstel, Amstelveen
  - Dialysecentrum Dianet (Amsterdam), Amsterdam
  - Reinier de Graaf Ziekenhuis, Delft
  - Deventer Ziekenhuis, Deventer
  - Catharina Ziekenhuis Eindhoven, Eindhoven
  - Maxima Medisch Centrum, Eindhoven
  - Martini Ziekenhuis, Groningen
  - Dialysecentrum Tergooi, Hilversum
  - Spaarne Gasthuis, Hoofddorp
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leiden UMC, Leiden
  - St. Jansdal ziekenhuis, Lelystad
  - Maastricht UMC+, Maastricht
  - St. Antonius Ziekenhuis, Nieuwegein
  - Radboud UMC, Nijmegen
  - Bravis ziekenhuis, Roosendaal
  - Franciscus Gasthuis en Vlietland, Rotterdam
  - Bernhoven, Uden
  - Diakonessenhuis Utrecht, Utrecht
  - Dialysecentrum Dianet (Utrecht), Utrecht
  - UMC Utrecht, Utrecht
  - VieCuri Medisch Centrum, Venlo
  - Isala Ziekenhuis, Zwolle
- Singapore General Hospital, Singapore, Singapore
- Spain (5):
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Arnau de Vilanova, Lleida
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Clinico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perkovic V, Jardine MJ, Neal B, Bompoint S, Heerspink HJL, Charytan DM, Edwards R, Agarwal R, Bakris G, Bull S, Cannon CP, Capuano G, Chu PL, de Zeeuw D, Greene T, Levin A, Pollock C, Wheeler DC, Yavin Y, Zhang H, Zinman B, Meininger G, Brenner BM, Mahaffey KW; CREDENCE Trial Investigators. Canagliflozin and Renal Outcomes in Type 2 Diabetes and Nephropathy. N Engl J Med. 2019 Jun 13;380(24):2295-2306. doi: 10.1056/NEJMoa1811744. Epub 2019 Apr 14. PMID 30990260
- [Background] Heerspink HJL, Jongs N, Chertow GM, Langkilde AM, McMurray JJV, Correa-Rotter R, Rossing P, Sjostrom CD, Stefansson BV, Toto RD, Wheeler DC, Greene T; DAPA-CKD Trial Committees and Investigators. Effect of dapagliflozin on the rate of decline in kidney function in patients with chronic kidney disease with and without type 2 diabetes: a prespecified analysis from the DAPA-CKD trial. Lancet Diabetes Endocrinol. 2021 Nov;9(11):743-754. doi: 10.1016/S2213-8587(21)00242-4. Epub 2021 Oct 4. PMID 34619108
- [Background] Chertow GM, Vart P, Jongs N, Toto RD, Gorriz JL, Hou FF, McMurray JJV, Correa-Rotter R, Rossing P, Sjostrom CD, Stefansson BV, Langkilde AM, Wheeler DC, Heerspink HJL; DAPA-CKD Trial Committees and Investigators. Effects of Dapagliflozin in Stage 4 Chronic Kidney Disease. J Am Soc Nephrol. 2021 Sep;32(9):2352-2361. doi: 10.1681/ASN.2021020167. Epub 2021 Jul 16. PMID 34272327
- [Background] Chewcharat A, Prasitlumkum N, Thongprayoon C, Bathini T, Medaura J, Vallabhajosyula S, Cheungpasitporn W. Efficacy and Safety of SGLT-2 Inhibitors for Treatment of Diabetes Mellitus among Kidney Transplant Patients: A Systematic Review and Meta-Analysis. Med Sci (Basel). 2020 Nov 17;8(4):47. doi: 10.3390/medsci8040047. PMID 33213078
- [Derived] Karsten M, Badve SV, Gansevoort RT, Berger SP, Heerspink HJL, Abrahams AC, Billot L, Bon RHACM, Gelens MACJ, Guinness D, Hamilton-Craig C, van Heerebeek L, Hemmelder MH, Houston L, Kozor R, Kuypers DRJ, Monaghan H, Neal B, Neuen BL, Otton J, Perkovic V, Rajwani A, Wang AY, Vervloet MG, Arnott C, Jakulj L; Renal Lifecycle Trial Cardiac Imaging Sub-studies Investigators. Cardiac impact of dapagliflozin in advanced chronic kidney disease: rationale and design of the Renal Lifecycle Trial cardiac imaging sub-studies. Clin Kidney J. 2025 Dec 2;19(1):sfaf376. doi: 10.1093/ckj/sfaf376. eCollection 2026 Jan. PMID 41551843
- [Derived] Garcia-Cosio Carmena MD, Farrero M, Blasco Peiro MT, Crespo M, Delgado Jimenez J, Diaz Molina B, Fernandez Rivera C, Garrido Bravo IP, Lopez Jimenez V, Melilli E, Mirabet Perez S, Perez Tamajon ML, Rangel Sousa D, Rodrigo E, Cruzado JM, Hernandez Marrero D; Spanish Society of Transplantation, the Spanish Society of Nephrology, and the Spanish Society of Cardiology (SET-SEC-SEN). Management of Kidney Disease in Heart Transplant Patients: A National Delphi Survey-based Consensus Expert Paper. Transplantation. 2025 Sep 1;109(9):e431-e445. doi: 10.1097/TP.0000000000005302. Epub 2025 Feb 7. PMID 39928546
- [Derived] Gill M, Leung M, Luo CY, Cheung C, Beauchesne A, Chang D, Lan J, Johnston O. Erythrocytosis and thrombotic events in kidney transplant recipients prescribed a sodium glucose cotransport-2 inhibitor. Clin Transplant. 2023 Aug;37(8):e15013. doi: 10.1111/ctr.15013. Epub 2023 May 11. PMID 37170711